CLINICAL TRIAL: NCT00799851
Title: Endoscopic Treatment of Esophageal Varices in Advanced Liver Disease Patients: a Randomized Controlled Trial Comparing Band Ligation and Cyanoacrylate Injection
Brief Title: A Randomized Controlled Trial Comparing Band Ligation and Cyanoacrylate Injection for Esophageal Varices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1244/04
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Liver Disease
Keywords: advanced liver disease; esophageal varices; band ligation; cyanoacrylate injection
MeSH Terms: conditions — Liver Diseases; Esophageal and Gastric Varices | interventions — Cyanoacrylates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Variceal band ligation (Active Comparator): VBL was performed with a multiband ligation device (Euroligator System®). The first band was placed at or close to the gastroesophageal junction, with subsequent bands being placed proximally in a slightly spiral pattern. All visible varices within the distal esophagus were treated, with a maximum of 10 bands being placed in each session. There was a 3-week interval between each treatment session. When VBL was technically impossible due to scarring, sclerotherapy with ethanolamine oleate was performed on thin vessels.
  Interventions: Device: Variceal band ligation
- cyanoacrylate injection (Active Comparator): CI group received intravariceal injections of 0.5 ml of N-butyl-2-cyanoacrylate (Histoacryl®) diluted in 0.5 ml of Lipiodol (Lipiodol®). Before injection of the Histoacryl-Lipiodol mixture, the catheter was filled up with 1 ml of Lipiodol. After puncturing the EV, the mixture was injected inside it and followed by injection of 1 ml of distilled water. Finally the catheter was retracted. To minimize the risk of embolism, a maximum of two medium or large vessels, in opposite walls, were treated in each session and not more than 0.5 ml of Histoacryl® was injected into each vessel.
  A second injection was performed in any EV that maintained blood flow (medium or large size, blue, depressive at palpation with the catheter), in a bi-weekly interval basis. A chest x-ray was performed to evaluate the location of the Histoacryl-Lipiodol solution. Small vessels were treated with ethanolamine oleate sclerotherapy.
  Interventions: Drug: cyanoacrylate injection

INTERVENTIONS:
Device: Variceal band ligation
  Arms: Variceal band ligation
Drug: cyanoacrylate injection — cyanoacrylate injection
  Arms: cyanoacrylate injection

SUMMARY:
Compare VBL and cyanoacrylate injection (CI) in the treatment of EV in patients with advanced liver disease regarding eradication, bleeding, mortality, complication and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* advanced liver disease (Child-Pugh ≥ 8 points)
* medium and/or large esophageal varices

Exclusion Criteria:

* prior endoscopic treatment.
* history of shunt operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-11; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Compare VBL and cyanoacrylate injection (CI) in the treatment of EV in patients with advanced liver disease regarding eradication, bleeding, mortality, complication and recurrence rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University Of São Paulo - Gastroenterology, São Paulo, São Paulo, Brazil